CLINICAL TRIAL: NCT05795920
Title: A Multicenter, One-arm Phase II Clinical Study of Utidelone Injection Combined With Gemcitabine in First-line Chemotherapy for Unresectable Advanced Pancreatic Cancer
Brief Title: Utidelone Injection Combined With Gemcitabine in First-line Chemotherapy for Unresectable Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTD1-PC-01
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: Unresectable advanced pancreatic cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced pancreatic cancer that is inoperable and not suitable for local treatment (Experimental): Patients with advanced pancreatic cancer that is inoperable and not suitable for local treatment
  Interventions: Drug: Utidelone injection in combination with gemcitabine

INTERVENTIONS:
Drug: Utidelone injection in combination with gemcitabine — Utidelone injection: 30mg/m2, for days 1-5, once a day, 21 days for a treatment week Period; Gemcitabine: 1000mg/m2, Q3W on day 1 and day 8, 21 days for a treatment cycle
  Other Names: UTD1

SUMMARY:
This trial is an efficacy and safety evaluation of the use of Utidelone injection in combination with gemcitabine for inoperable and locally inappropriate use first-line chemotherapy in the treatment of advanced pancreatic cancer.

Main Purpose:To evaluate the use of utidelone in combination with gemcitabine in unresectable, advanced pancreatic cancer without progressionSurvival (PFS), overall survival (OS), duration of response (DOR), and safety; Secondary objective: Use of utidelone in combination with gemcitabine in patients with unresectable, advanced pancreatic cancer, according to investigators Objective response rates (ORRs) assessed against RECIST v1.1 criteria.

DETAILED DESCRIPTION:
This trial is a multicenter, single-arm phase II clinical trial of Utidelone (UTD1) injection combined with gemcitabine in patients with unresectable, advanced pancreatic cancer, and the study will include 6 centers and enroll 92 patients.Patients who met the entry criteria received Utidelone in combination with gemcitabine: Utidelone (utidelone ®) injection: 30 mg/m2, administered daily on Days 1-5, in 21-day cycles; gemcitabine: 1000 mg/m2, administered 3 weeks using (Q3W) on Days 1 and 8, in 21-day cycles; treatment period: 6-8 cycles, or until the patient experienced disease progression or intolerable toxicity or death.Tumor assessments will be performed at baseline and every 6 weeks (± 7 days) after enrollment until disease progression according to response evaluation criteria in solid tumours (RECISTv1.1) criteria.For patients without disease progression, tumor assessments will continue regardless of whether or not the patient discontinues study treatment unless consent is withdrawn.Follow-up data collection, including subsequent anticancer therapy, was to occur until patient death, withdrawal of consent, loss to follow-up, or study termination, whichever came first.Safety assessments assessed the incidence, nature, and severity of adverse events and laboratory abnormalities according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 in the Investigator-Initiated Clinical Trial (IIT) Study UTD1-PC-01 14 in Shanghai First People 's Hospital.Laboratory safety assessments included periodic monitoring of hematology and chemistry.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the study must meet all of the following criteria:

1. Age: 18-75 years old.
2. Karnofsky (KPS) physical status score ≥70.
3. Those confirmed by histopathology or cytology, inoperable and unsuitable for local treatment This is a malignant tumor of pancreatic ductal epithelium, graded as stage Ⅲ-Ⅳ according to the American Joint Committee on Cancer (AJCC) eighth Edition (T4NxM0-1/TxNxM1), except for pancreatic neuroendocrine tumors;
4. Baseline blood routine and biochemical indexes of subjects meet the following standards: hemoglobin ≥90g/L; neutral Granulocyte absolute count (ANC) ≥1.5×109g/L; Platelet ≥100×109/L; glutamine Enzyme (ALT), aspartate aminotransferase (AST) ≤2.5 times the normal upper limit; Serum total bilirubin <1.5 times the normal upper limit; Serum creatinine <1 times the normal upper limit; Serum albumin

   ≥30g/L.
5. Cardiac function: a) left ventricular ejection fraction (LVEF) ≥50%; b) 12-ECG showed no myocardial ischemia; c) No history of arrhythmia requiring drug intervention before enrollment;
6. No severe concomitant disease with survival time <5 years, known peripheral nerve disease ≤ grade 1.
7. Agree to and be able to follow the protocol during the study.
8. Provide written informed consent before entering the study screening. -

Exclusion Criteria:

1. For patients with pancreatic cancer who had previously received chemotherapy, radiotherapy or immunotherapy.
2. Patients with pancreatic neuroendocrine tumors confirmed by histopathology or cytology
3. Pregnant or lactating women.
4. Women of childbearing age who had a positive pregnancy test at baseline or did not undergo a pregnancy test. Postmenopausal women must Stop menstruation for at least 12 months before pregnancy is not possible.
5. Men and women who had sex (with the possibility of procreation) were reluctant to use contraception during the study period.
6. Non-melanoma skin cancer and cervical carcinoma in situ were cured in patients with other malignant history in the last 5 years Outside.
7. A history of uncontrolled epilepsy, central nervous system disease or mental disorder, as determined by the investigator Clinical severity can prevent the signing of informed consent or affect patient adherence to oral medication.
8. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, New York Heart Association May have grade II or worse congestive heart failure or severe cardiac rhythm requiring medical intervention Disorder, or history of myocardial infarction within the last 12 months.
9. Those who are severely allergic to polyoxyethylene (35) castor oil, or have used anti-microtubule drugs in the past Severe adverse reactions occurred.
10. Known peripheral nerve disease ≥NCICTC, AE grade 2.
11. severe uncontrolled recurrent infection, or other severe uncontrolled concomitant disease.
12. Moderate or severe renal impairment [creatinine clearance ≤50ml/min (according to Cockrcoft and Gault equation), or serum creatinine > upper normal limit (ULN) .
13. Acute or chronic active hepatitis B, hepatitis C infection, hepatitis B virus (HBV) DNA > 2000 IU/ml or 104 copies /ml, Hepatitis C virus (HCV) RNA > 103 copies /ml, hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive at the same time, human immunity Epidemic defect virus (HIV).
14. Allergic to Utidelone or gemcitabine.
15. Participants who had received study medication or preparation/treatment (i.e., participating in other trials) within 4 weeks prior to enrollment.
16. Patients who were not eligible to participate in the study for any reason determined by the investigator.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-07-08 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause assessed up to 100 months
  Time from enrollment to death (from any cause)
progression free survival progression free survival | From date of randomization until the date of first documented progression assessed up to 100 months
  Disease progression from baseline assessment of enrollment to first radiographically verifiable disease progression (PD) (RECIST 1.1 standard) or deaths from any cause where progression was not recorded Time.

SECONDARY OUTCOMES:
Duration of response Duration of Response | Time from complete response/partial response (CR/PR) to progression/death (from any cause), assessed up to 100 months
  That is, from the first time the evaluation results meet CR or PR criteria to the observation of PD or death

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, Prof., Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No